CLINICAL TRIAL: NCT00361699
Title: Effect of 3-hydroxy-3-methylglutaryl-coenzyme A(HMG-CoA) Reductase Inhibitor Upon the Serum High Sensitive CRP in the Post-ischemic Patients With Hyperlipidemia During the Prospective Study of J-STARS.
Brief Title: hsCRP in Japan Statin Treatment Against Recurrent Stroke (J-STARS hsCRP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government); Hiroshima University (Other); Osaka University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: J-STARS hsCRP; C000000211 (Other: UMIN CTR)
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Ischemic Stroke
Keywords: stroke; brain ischemia; cerebrovascular accident; statin; hydroxymethylglutaryl-CoA reductase inhibitors; cholesterol; hypercholesterolemia; hyperlipidemia; multicenter studies; prospective studies; endpoint determination; randomized controlled trials; recurrence; pravastatin; c-reactive Protein
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Ischemia; Hypercholesterolemia; Hyperlipidemias; Recurrence | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

ARMS (2):
- Pravastatin (Active Comparator): Patient has 10mg oral administration of Pravastatin per day. It starts within one month from their entry and continues every day until the end of the study or its endpoints.
  Interventions: Drug: Statin
- No intervention (No Intervention): Patient has no intervention.

INTERVENTIONS:
Drug: Statin
  Arms: Pravastatin

SUMMARY:
Inhibition of 3-hydroxy-3-methylglutaryl-coenzyme A(HMG-CoA) reductase can play a role in preventing recurrent vascular events from ischemic heart disease patients, whose mechanism consists in not only the reduction of serum lipid level but also anti-inflammatory effects. Serum high sensitive CRP is known to be a predictor of cardiovascular events independent of other conventional risk factors. The present substudy examine whether such pleiotrophic effect of HMG-CoA reductase inhibitor (statin) which decreases high sensitive CRP would be observed in the post-ischemic stroke patients who have already been registered in the J-STARS, and the relationship the values of high sensitive CRP and recurrence of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke except for cardiogenic embolism, from 1 month to 3 years after onset
* Hyperlipidemia and total cholesterol level of 180-240mg/dl without the prescription of statin within previous 30 days
* Able to visit outpatient department
* Informed consent on the form filled in by the patient.

Exclusion Criteria:

* Ischemic stroke of other determined cause according to the TOAST classification
* Ischemic heart disease and necessary to use statin
* Hemorrhagic disorders
* Platelet count <=100,000/ul within 3 months prior to study start
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>= 100IU/L within 3 months prior to study start
* Serum creatinine >=2.0mg/dl within 3 months prior to study start
* A scheduled operation
* The presence of malignant disorder

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 2004-03; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
serum level of high sensitive CRP | until the last day of the next February after 5-year follow-up survey

SECONDARY OUTCOMES:
recurrent stroke | until the last day of the next February after 5-year follow-up survey

CONTACTS AND LOCATIONS:
Overall Officials: Masayasu Matsumoto, MD, PhD, Principal Investigator — Hiroshima University Hospital
Locations (2):
- Japan (2):
  - Hiroshima University Hospital, Hiroashima, Hiroshima
  - Osaka University, Suita-shi, Osaka

REFERENCES:
- See also: Available only in Japanese — http://jstars.umin.ne.jp